CLINICAL TRIAL: NCT01540617
Title: The Neural Basis of Lumbosacral Proprioceptive Impairment in Recurrent Low Back Pain
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Prof. dr., KU Leuven
Other Study IDs: 2012_SBrumagne_MRIproprio
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Low Back Pain
Keywords: Low back pain; Proprioception; Postural control; Spine; Variability; MRI; Vibration; Brain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Persons with low back pain
- Healthy persons

SUMMARY:
Low back pain (LBP) is a well known health problem in Western society that is significantly responsible for socio-economic problems like absenteeism and disability. The lifetime prevalence of LBP is 60-80% and approximately 85% of this LBP has a "non-specific" character whereby the underlying causes and risk factors cannot be demonstrated. While many people recover within a month, most individuals will have recurrence within a year with more severe symptoms. This might be due to insufficient knowledge of the underlying mechanisms. Impaired proprioception, the ability to discern body/limb positions and movements, may cause and maintain LBP shown by an altered postural control strategy. Specifically, patients with LBP rely more on proprioceptive signals from the ankles due to less reliable proprioceptive input of proximal segments. Moreover, they show a decreased variability in postural control and less postural robustness, while variability is a prerequisite for optimal functioning of biological systems. However, further clarification of the neural correlates is necessary. Deficits in proprioception, as found in a subgroup of patient with LBP, are associated with a decreased ability of the brain to process proprioceptive inputs.

The aim of this project is to clarify the central changes in individuals with recurrent non-specific low back pain and healthy controls. To evaluate these central changes MRI techniques (3DTFE, DTI and RS-fMRI) will be used. In addition, the association between central changes and postural control tasks will be evaluated.

ELIGIBILITY:
Inclusion Criteria persons with low back pain:

* Age: 20-50 year
* At least 6 months of low back pain with/without referred pain in buttock/thigh
* At least 3 episodes of disabling low back pain
* At least a score of 14% on the Oswestry Disability Index
* Willingness to sign the informed consent
* Met the MRI related requirements

Inclusion Criteria healthy persons:

* Age: 20-50 year
* No history of low back pain
* A score of 0% on the Oswestry Disability Index
* Willingness to sign the informed consent
* Met the MRI related requirements

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson, MS, Stroke with sequels....
* Radicular symptoms
* Not Dutch-speaking
* Strong opioids
* Neck pain
* Ankle problems
* Smoking

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Leuven and surrounding area
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Structural changes in white matter pathways (3DTFE and DTI) (in individuals with recurrent non-specific low back pain compared to healthy controls) | One time point
Changes in resting state activity between individuals with recurrent non-specific low back pain and healthy controls) | One time point
Proprioceptive postural control (center of pressure displacement in response to muscle vibration) | One time point

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, Professor, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

REFERENCES:
- [Background] Claeys K, Brumagne S, Dankaerts W, Kiers H, Janssens L. Decreased variability in postural control strategies in young people with non-specific low back pain is associated with altered proprioceptive reweighting. Eur J Appl Physiol. 2011 Jan;111(1):115-23. doi: 10.1007/s00421-010-1637-x. Epub 2010 Sep 8. PMID 20824281
- [Background] Brumagne S, Janssens L, Knapen S, Claeys K, Suuden-Johanson E. Persons with recurrent low back pain exhibit a rigid postural control strategy. Eur Spine J. 2008 Sep;17(9):1177-84. doi: 10.1007/s00586-008-0709-7. Epub 2008 Jul 2. PMID 18594876
- [Background] Brumagne S, Janssens L, Janssens E, Goddyn L. Altered postural control in anticipation of postural instability in persons with recurrent low back pain. Gait Posture. 2008 Nov;28(4):657-62. doi: 10.1016/j.gaitpost.2008.04.015. Epub 2008 Jun 9. PMID 18541428